CLINICAL TRIAL: NCT01804751
Title: Prediction of Adverse Perinatal Outcome for Preeclampsia in Sichuan Province of China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: West China Second University Hospital (Other)
Collaborators: Sichuan Academy of Medical Sciences (Other); Guang'an people's hospital of Sichuan province (Other); The First People's Hospital of Neijiang (Other); Suining Central Hospital (Other); Sichuan Provincial Maternal and Child Health Care Hospital (Unknown); Chengdu Women's and Children's Central Hospital (Other); Luzhou Medical College (Other); pengzhou shi fuyou baojianyuan (Unknown); Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Xinghui Liu, professor, West China Second University Hospital
Other Study IDs: hx2ck2
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2013-06

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to build a model for the prediction of adverse perinatal outcome for preeclampsia in china

ELIGIBILITY:
Inclusion Criteria:

* admitted with preeclampsia or had developed preeclampsia after admission

Exclusion Criteria:

* admitted in spontaneous labour or had achieved any component of the maternal outcome before either fulfilling eligibility criteria or collection of predictor data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese women who fulﬁlled a research deﬁnition of preeclampsia, and who were admitted to participating obstetric centres
Sampling Method: Non-Probability Sample
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
maternal mortality | within 48h of eligibility

SECONDARY OUTCOMES:
serious central nervous system morbidity | within 48h of eligibility
serious cardiorespiratory morbidity | within 48h of eligibility
serious hepatic morbidity. | within 48h of eligibility
serious renal morbidity | within 48h of eligibility
serious haematological morbidity | within 48h of eligibility